CLINICAL TRIAL: NCT05481060
Title: The Effect of Screen-based Simulation Method on the Attitudes and Practices of Nursing Students on Intimate Partner Violence
Brief Title: The Attitudes and Practices of Nursing Students on Intimate Partner Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gamze Agartioglu Kundakci, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 714
Record Dates: First submitted 2022-07-18; First posted 2022-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Nursing Students
Keywords: intimate partner violence; nursing student; screen-based simulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screen-based simulation (Experimental): Screen-based simulation about intimate partner violence against women prepared by researchers will apply to nursing students.
  Interventions: Other: Screen-based simulation
- Control group (No Intervention): Online didactic education about intimate partner violence against women prepared by researchers will apply to nursing students.

INTERVENTIONS:
Other: Screen-based simulation — In the research, training will be given to the experiment group on intimate partner violence against women through screen-based simulation.
  Arms: Screen-based simulation

SUMMARY:
The purpose of this research is to determine the effect of screen-based simulation method on nursing students' attitudes and practices about intimate partner violence against women.

DETAILED DESCRIPTION:
Intimate partner violence (ipv) against women is characterized as a global epidemic in health care delivery due to its prevalence, high morbidity, and mortality. One of the first healthcare providers that victims interact with is nurses. Nurses should have sufficient knowledge and skills to fulfill their roles and responsibilities defined in the issue of ipv against women. Educational environments must provide nursing students with the opportunity to be aware of ipv against women and to manage cases. Institutions that add simulation content to their education programs have the potential to become the gold standard when preparing nursing students for case management of ipv against women. Screen-based simulations (SBSs) use available digital technology to represent patients, populations, or other healthcare encounters on a computer screen or a mobile tablet, smartphone, or other screen-based devices. Simulations using screens have advantages over mannequin-based simulations-the software is infinitely replicable, the simulation programs can be portable, they can be accessed asynchronously without a live instructor present, and the software can be distributed to many devices, and the programming can track massive amounts of usage data. The purpose of this research is to determine the effect of screen-based simulation method on nursing students' attitudes and practices about intimate partner violence against women. The intervention and control groups of the study with the pre-test, post-test randomized controlled experimental design will comprise fourth-year students attending a university's nursing faculty. Power analysis was performed to calculate the sample size and it was planned to include 63 students in the sample group. In the research, the intervention group will be trained on ipv through SBSs whereas the control group will be trained via online conference. The research outputs will be measured by Health Workers' Attitudes and Practices on Intimate Partner Violence Against Women Scale, Simulation Design Scale and Debriefing Experience Scale.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being a 4th-year student in the nursing department

Exclusion Criteria:

* Having worked as a nurse before
* To have taken an elective course on violence against women in undergraduate education
* To be married

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
The Attitudes and Practices of Healthcare Providers Regarding Intimate Partner Violence (APHCPs-IPV) survey scale | Before the recruit pre-test (APHCPs-IPV survey scale) will be applied. Six months after the intervention post-test (APHCPs-IPV survey scale) again will be applied. Researchers will measure change from APHCPs-IPV survey scale at 6 months.
  The Turkish version of the scale of 42 items and consists of eight subscales. The subscales are (a) preparedness, (b) self-confidence of the practitioner, (c) lack of control, (d) comfort following disclosure, (e) professional support, (f) practice pressures, (g) abuse inquiries, and (h) practitioner consequences of asking. It is scored on a 4-point scale ranging from 1 to 4 (1- strongly agree, 2 agree, 3-disagree, and 4-strongly disagree). The APHCPs-IPV scale total scores range from 42 to 168. Higher scores reflected greater self-reported preparedness, self-confidence, feelings of professional support, comfort with abuse inquiries, and comfort with discussions following disclosure as well as decreased concern about the consequences of abuse inquiries and decreased feelings of no control and system pressures.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No